CLINICAL TRIAL: NCT01139333
Title: Evaluation of Mer and Axl Expression in Acute Myeloid Leukemia Patient Samples
Brief Title: Blood and Tumor Tissue Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B4; COG-AAML10B4 (Other: Children's Oncology Group); CDR0000671452 (Other: Clinical Trials.gov); NCI-2011-02222 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-05; First posted 2010-06-08 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Blotting, Western; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood and tumor samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: western blotting
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying blood and tumor tissue samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate Mer and Axl expression in samples from pediatric patients with acute myeloid leukemia (AML).
* To determine if abnormal expression of Mer and Axl is associated with poor clinical characteristics (e.g., induction failure or relapse) of AML in these patients.

OUTLINE: This is a multicenter study.

Archived samples from pediatric patients with acute myeloid leukemia are analyzed for Mer and Axl expression by flow cytometry and western blot assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Children Oncology Group (COG) patient samples

PATIENT CHARACTERISTICS:

* Available clinical data

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2009-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Expression of Mer and Axl
Association of abnormal expression of Mer and Axl with induction failure or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M. Eisenman, MD, Principal Investigator — University of Colorado, Denver